CLINICAL TRIAL: NCT01156870
Title: Dose Escalation, Safety and Pharmacokinetic, First in Man Study, of SAR566658 Administered as a Single Agent by Intravenous Infusion in Adult Patients With CA6-Positive and Refractory Solid Tumors
Brief Title: First in Man Study of SAR566658 Administered in Patients With CA6-Positive and Refractory Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED10499; U1111-1116-4129 (Other: UTN)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — SAR-566658

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR566658 (Experimental): SAR566658 will be administered by intravenous (IV) infusion according to three different schedules
  Interventions: Drug: SAR566658

INTERVENTIONS:
Drug: SAR566658 — Pharmaceutical form:solution for infusion
  Route of administration: intravenous

SUMMARY:
Primary Objective:

To determine the maximum tolerated dose (MTD) of SAR566658

Secondary Objectives:

* To characterize the safety profile of SAR566658
* To evaluate the pharmacokinetic profile of SAR566658
* To assess the potential immunogenicity of SAR566658
* To assess preliminary antitumor activity
* To assess the effect of SAR566658 at recommended dose on CYP3A enzyme activity using midazolam
* To assess safety in the alternative schedules of SAR566658 administration

DETAILED DESCRIPTION:
The duration of the study for one patient in the dose escalation phase of the study will include a screening period of up to 3 weeks, a 3-week treatment cycle(s) and a 2-week treatment cycle(s). The patients may continue treatment until disease progression, unacceptable toxicity, or willingness to stop, followed by a minimum of 30-day follow-up. If a patient treated in dose escalation part or in an expansion cohorts, continues to benefit from the treatment at the time of Clinical Study Report, the patient can continue study treatment and will continue to undergo all assessments as per the study flowchart. Such patients will be followed at least until 30 days after the last IMP administration.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of CA6-positive solid tumors as moderate to intense membrane staining of ≥15% of tumor cells for which no standard therapy is available.

Exclusion criteria:

* Eastem Cooperative Oncology Group performance status ≥2.
* Any serious active disease or co-morbid condition, which, in the opinion of the Investigator, may interfere with the safety or the compliance with the study.
* Poor bone marrow reserve.
* Poor liver and renal function.
* Pregnant or breast-feeding woman.
* No use of effective birth control methods, when applicable.
* No resolution of all specific toxicities (excluding alopecia) related to any prior anti-cancer therapy to Grade ≤1 according to the National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.03 grade scaling.
* Wash out period of less than 3 weeks from previous antitumor therapy or any investigational treatment, (and less than 6 weeks in case of prior nitroso-urea and or mitomycin C treatment). Patients will be eligible if hormonotherapy (ie, for breast tumors) is discontinued before first Investigational product administration.
* Wash out period of less than 1 week from last palliative dose of radiotherapy.
* Patients with respiratory insufficiency defined by a decrease more than 50% compared to theoretical baseline pulmonary volumes and theoretical baseline Diffusing capacity of the Lung for Carbon monoxyde.
* Any lung radiotherapy in patient's cancer history.
* Patients with previous history or active interstitial lung disease or pulmonary fibrosis.
* Patients with abnormal cardiac function defined by a Left Ventricular Ejection Fraction <50%.
* Patients with previous history of acute cardiac failure.
* Patients with previous history and/or unresolved corneal disorders.
* Known intolerance to infused protein products or maytansinoids.
* Patients treated with strong CYP3A inhibitors within 2 weeks prior study drug administration.
* For patients to be treated in the midazolam cohort:
* Any treatment known to induce CYP3A isoenzymes or to inhibit CYP3A4 activities not allowed within 2 weeks before midazolam administration and up to the end of pharmacokinetic sampling following the last midazolam administration.
* Any contra-indications to midazolam, according to the applicable labeling.
* Patients older than 60 years.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Dose Escalation to determine the maximum tolerated dose (MTD) of SAR566658 | 3 weeks
Extension Cohorts to evaluate the preliminary anti-tumoral effect of SAR566658 | Anticancer activity is assessed every 6 weeks
To assess the effect of SAR566658 at the recommended dose on CYP3A enzyme activity using midazolam as probe | At D1 and D4 of administration of SAR566658 for 24h of midazolam dosing

SECONDARY OUTCOMES:
Overall safety profile based on adverse events reporting, laboratory tests, vital signs and specific pulmonary and ocular tests, according to the NCI-CTC AE v4.03 | Up to 2 years
Pharmacokinetic (PK) parameters | Up to 2 years
Immunogenicity evaluation (anti-drug antibodies) | Up to 2 years
Antitumoral response | Up to treatment discontinuation
To assess the effect of SAR566658 at recommended dose on CYP3A enzyme activity using midazolam | Up to Cycle 2
To assess safety in the alternative schedules of SAR566658 administration | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- United States (2):
  - Investigational Site Number 840002, Cincinnati, Ohio
  - Investigational Site Number 840001, San Antonio, Texas
- Investigational Site Number 250001, Toulouse, France
- Spain (2):
  - Investigational Site Number 724002, Madrid
  - Investigational Site Number 724001, Madrid